CLINICAL TRIAL: NCT05006924
Title: Symptoms and Outcome Measures for Upper- Limb Function in Myotonic Dystrophy Type 1
Acronym: SOUL-DM1
Status: Completed | Type: Observational
Sponsor: Oslo University Hospital (Other)
Collaborators: University of Oslo (Other); Haukeland University Hospital (Other)
Responsible Party: Principal Investigator, Kristin Ørstavik, PI, Oslo University Hospital
Other Study IDs: 255164
Record Dates: First submitted 2021-08-10; First posted 2021-08-16 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Myotonic Dystrophy 1
Keywords: Outcome measure; Patient reported outcome; Upper limb function; arm- and hand function; Symptoms
MeSH Terms: conditions — Myotonic Dystrophy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Myotonic Dystrophy type 1 (DM1) is a multisystem disease that causes muscle weakness and myotonia. As a result upper limb function might become impaired. In this study we will examine patients with DM1 and record their upper limb function. We will will use a battery of patient reported outcomes (PROs) and Outcome measures (OMs) in order to evalute which ones are suitable for use in clinical practise and research studies.

ELIGIBILITY:
Inclusion Criteria:

• Genetically confirmed Myotonic Dystrophy type 1

Exclusion Criteria:

* Unable to answer or understand questionnaires due to language barriers or cognitive status
* Unable to perform functional tests

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with Myotonic Dystrophy type 1 in Norway
Sampling Method: Non-Probability Sample
Enrollment: 89 (Actual)
Dates: Start 2021-12-10 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
Motor Function Measures (MFM) | 30-45 minutes
  Functional test
Nine Hole Peg Test | 1-3 minutes
  Fine motor function test
Myogrip/Dynamometer | 1-3 minutes
  Measures hand strenght
Myopinch | 1-3 minutes
  Measures finger strenght
ABILHAND Questionnaire | 5 min
  A measure of manual ability for adults with upper limb impairments. The scale measures a person's ability to manage daily activities that require the use of the upper limbs, whatever the strategies involved. Consists of 22 questions (18 to be answered by adults). The categories are easy, difficult or unable to perform. The querionnaire gives a sum score where higher score equals better function.Score from 0 to 36
ACTIVLIM Questionnaire | 5 min
  A measure of activity limitations for patients with upper and/or lower limb impairments. The scale measures a patient's ability to perform daily activities requiring the use of the upper and/or the lower limbs, whatever the strategies involved. Consists of 22 questions (18 to be answered by adults). The categories are easy, difficult or unable to perform. The questionnaire gives a sum score where higher score equals better function. Score fror 0 to 36

SECONDARY OUTCOMES:
Trunk Impairment Scale - modified Norwegian version | 8-15 minutes
  Motor impairment of trunk measured by functional testing. Six subdomains measuring stability and mobility of trunkal movement. Min score 0 - Max score 16. Higher score indicates better function.
Four Square Step Test | 1-3 minutes
  Dynamic balance test
PROMIS29 | 5-10 minutes
  This a compostie measurement that is a Questionnaire. Patient reported outcome measure. Generic health related quality of life assesses each of the 7 PROMIS domains (depresseion, anxiety, physical function, pain, fatigue, sleep disturbance and ability to participate in social roles). The PROMIS 29 questionnaire contains 4 questions from each of seven PROMIS contents (physical function, depression, anxiety, fatigue, sleep disorder, participation in social activities and pain interaction) and 1 question from the intensity of pain. Each item has 5 answer options (from 1 to 5), only pain intensity has 11 answer options (from 0 to 10). From the sum of the answers to each question in the domain, the total raw score for each domain is calculated, resulting in seven domain scores, each between 4 and 20.
Starkstein Apathy Scale | 5 minutes
  Questionnaire to be filled in under guidance of interviewer. Patient reported outcome measure of apathy. 14 questions, each of which is scored on a 4-point scale of 0-3, and apathy is rated as severer as the total score (0-42) increases
Montreal Cognitive Assessment (MoCA) | 10 minutes
  Cognitive assessment screening questionnaire. To be filled out in an interview setting. Score from 0 to 30, where a higher score indicates a better cognitive function. A score of 26 or more is considered normal.
Lung function test | 10 minutes
  Spirometry with FVC (Forced Vital Capasity)
Lung function test | 10 minutes
  PEF (Peak Expiratory Flow).

CONTACTS AND LOCATIONS:
Overall Officials: Kristin L Ørstavik, PHD, Principal Investigator — Oslo University Hospital; Hilde S Robinson, PHD, Study Director — University of Oslo
Locations (3):
- Norway (3):
  - Haukeland University Hospital, Bergen
  - Oslo University Hispital, Oslo
  - Frambu Centre for Rare Disorders, Siggerud

IPD SHARING:
Plan to Share IPD: No